CLINICAL TRIAL: NCT02834351
Title: Atteinte Tissulaire au Cours de l'ischémie Chronique d'Effort. Validation d'un modèle d'étude du Muscle Sartorius Humain
Brief Title: Tissue Lesions in Exercise Related Ischemia
Acronym: SARTORIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013-A00166-39
Record Dates: First submitted 2016-06-16; First posted 2016-07-15 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Ischemia; Peripheral Artery Disease
MeSH Terms: conditions — Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peripheral artery diseased group (Active Comparator): pad Patients referred for femoro popliteal bypass Muscle biopsy during surgery
  Interventions: Other: Muscle Biopsy
- Cardiac group (Sham Comparator): Patients referred for saphenous withdrawal for coronary bypass Muscle biopsy during surgery
  Interventions: Other: Muscle Biopsy

INTERVENTIONS:
Other: Muscle Biopsy — A distal and proximal biopsy of the sartorius muscles ( 0.5 cm3 each) will be performed during surgery for saphenous vein withdrawal (cardiac group) or arterial bypass (PAD group) The samples are then treated with neurovascular and mitochondrial biology laboratory.
  the activity of the complex 1 is analyzed and compared between the 2 groups.

SUMMARY:
The purpose of this study is to evaluate the effect of muscle ischemia during claudication on mitochondrial function.

Comparison to patients with arterial disease but absence of lower limb claudication (Cardiac group) feasibility study.

DETAILED DESCRIPTION:
Assess the feasibility of the study of micro-vascular function and mitochondrial on muscle sample (sartorius) in a group of arterial disease and non arteriopathy group.

Analysis of the activity of mitochondrial chain Immunochemistry of tissue markers

ELIGIBILITY:
Inclusion Criteria:

* Intervention for femoropopliteal bypass (PAD group)
* Intervention for saphenous withdrawal for coronary bypass surgery (cardiac group)

Exclusion Criteria:

* Participate in another biomedical research
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Activity differences in mitochondrial complex I between the distal and proximal levy in group 1 and group 2. | 1 week
  Measurement of mitochondrial complex 1 activity (arbitrary units) on muscle biopsies by the laboratory of biochemistry. Comparison of the results observed on the same miuscle at the proximal level (assumed normal in both groups) and distal level (assumed ischemic in claudicants but not in cardiac patients without limb symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, PROFESSOR, Principal Investigator — UH ANGERS
Locations (1):
- Uh Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No